CLINICAL TRIAL: NCT01319318
Title: Observational Study of Ocular Inflammation in Patients Undergoing a Pars Plana Vitrectomy
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-OZU-10-017
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-04

CONDITIONS: Vitrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pars Plana Vitrectomy: Pars plana vitrectomy performed in study eye on Day 0.
  Interventions: Procedure: Pars Plana Vitrectomy

INTERVENTIONS:
Procedure: Pars Plana Vitrectomy — Pars plana vitrectomy performed in study eye on Day 0.

SUMMARY:
This study will evaluate the degree of post-operative ocular inflammation in patients who are undergoing a pars plana vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Require pars plana vitrectomy in at least 1 eye
* Best corrected visual acuity in the study eye between 20/400 and 20/40

Exclusion Criteria:

* Use of any NSAIDs (topical or systemic) within 14 days
* Use of topical or systemic steroids within 30 days
* Active eye infection in either eye
* Any eye surgery within 6 months
* Prior pars plana vitrectomy, YAG capsulotomy or uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who plan on undergoing a pars plana vitrectomy
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pars Plana Vitrectomy
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pars Plana Vitrectomy
Number analyzed (Participants) | 25
Age Continuous [Mean (Standard Deviation); unit: Years] | 69.6 (10.06) [47 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Vitreous Cell Count of 0
Description: The study eye was dilated and the investigator used an instrument to count the number of visible cells in the vitreous, the jelly-like fluid that fills the back of the eye, using the following scale: 0 (no cells) best, +1 (1-10 cells), +2 (11-30 cells), +3 (31-50 cells) and +4 (>50 cells) worst.
Time Frame: Week 4
Population: Intent to treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Pars Plana Vitrectomy
Number analyzed (Participants) | 25
Percentage of participants | 88.0

ADVERSE EVENTS:
Arm/Group | Pars Plana Vitrectomy
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pars Plana Vitrectomy (N=25)
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pars Plana Vitrectomy (N=25)
Ocular pain (Eye disorders) | 9
Eye redness (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.